CLINICAL TRIAL: NCT00038025
Title: A Phase II Study of Deoxycoformycin (DCF) in Lymphoid Malignancies
Brief Title: A Study Of Deoxycoformycin(DCF)/Pentostatin In Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM94-026
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Mycosis Fungoides; Lymphoma; Chronic lymphocytic leukemia; Deoxycoformycin; Pentostatin; All other lymphomas; Nucleoside analogue; Adenosine deaminase inhibitor; T-cells
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Leukemia, Lymphocytic, Chronic, B-Cell; Mycosis Fungoides; Lymphoma | interventions — Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deoxycoformycin (DCF)/Pentostatin (Experimental)
  Interventions: Drug: Deoxycoformycin (DCF)

INTERVENTIONS:
Drug: Deoxycoformycin (DCF) — Patients received Deoxycoformycin (DCF)/Pentostatin administered by intravenous bolus daily over a consecutive 3-day period. This course was repeated at 3-week intervals.
  Other Names: Nipent; Pentostatin

SUMMARY:
The purpose of this study is to determine the side effects and antitumor response of patients with lymphoid malignancies to Deoxycoformycin (DCF)/Pentostatin.

DETAILED DESCRIPTION:
Deoxycoformycin(DCF)/Pentostatin is a T-cell cytotoxic drug with previously reported responses in lymphoid malignancies but larger studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of lymphoid malignancy with an expected complete response rate of less than 20 percent OR have failed at least one prior therapy.
* No chemotherapy within 3 weeks of entry into study and must have recovered from acute toxic effects of prior therapy.
* Life expectancy of at least 12 weeks.
* Performance status equal to or less than Zubrod 2.
* Signed informed consent.
* Patients with measurable disease.
* Age at least 16 years.
* Adequate bone marrow function (unless involvement of bone marrow by lymphoma) defined as AGC greater than 1500 and platelet count greater than 100,000.
* Adequate hepatic function with a bilirubin less than or equal to 1.5 mg % and SGPT less than or equal to 4 times the upper limits of normal.
* Adequate renal function defined as serum creatine less than or equal to 1.5 mg %.

Exclusion Criteria:

* No serious intercurrent illness.
* Adequate contraception (if applicable).
* NO patients with significant cardiac disease, i.e. New York Heart Association (NYHA) class III or IV.
* NO experimental clinical trial within 3 weeks of study entry.
* NO patients with active CNS disease.
* Full recovery from any prior surgical treatment.
* NO active active infections.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1994-09-06 (Actual); Primary Completion 2006-11-29 (Actual); Study Completion 2006-11-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Overall Response | Baseline and approximately every 3 weeks thereafter
  Overall responses (OR) of participants with lymphoid malignancies to Deoxycoformycin (DCF)/Pentostatin defined as Complete Response (CR) and Partial Response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Principal Investigator — MD Anderson
Locations (1):
- M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Public website for M. D. Anderson Cancer Center — http://www.mdanderson.org